CLINICAL TRIAL: NCT05962476
Title: Transcutaneous Vibro-Acoustic Therapy in Parkinson Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study discontinued due to a lack of resources.
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Prabesh Kanel, Research Investigator, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00231771
Record Dates: First submitted 2023-06-29; First posted 2023-07-27 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Parkinson Disease
Keywords: transcutaneous vibro-acoustic therapy; anxiety
MeSH Terms: conditions — Parkinson Disease; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Parkinson's Disease (Experimental): Participants will use the vibro-acoustic device 90-120 days for 6 hours at night on the Apollo Neuro setting "Sleep and Renew".
  Interventions: Device: Transcutaneous vibro-acoustic device

INTERVENTIONS:
Device: Transcutaneous vibro-acoustic device — Wearable device which sends low-frequency sound vibrations through the skin.
  Other Names: Apollo Neuro

SUMMARY:
Small exploratory pilot study to assess effects of a transcutaneous vibro-acoustic therapy device (Apollo Neuro) in people with Parkinson's disease (PD).

DETAILED DESCRIPTION:
The overarching goal of this study is to investigate changes in anxiety, nighttime heart rate variability, and fear of falling in people with PD before and after 3-months usage of a transcutaneous vibro-acoustic therapy device. Positive findings in this small exploratory pilot trial may support future studies of transcutaneous vibro-acoustic therapy for individuals with PD.

This study was terminated due to lack of resources. One participant was consented, but no data was collected.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Parkinson's Disease (Hoehn and Yahr stage 2 or higher)
* Individuals on or off dopaminergic therapy
* Present of anxiety or panic disorder
* Fear of falling
* Understanding of use and care of smart phones and devices

Exclusion Criteria:

* Presence of significant dementia
* Disorders which may resemble PD, such as dementia with Lewy bodies, vascular dementia, normal pressure hydrocephalus, multiple system atrophy, corticobasal ganglionic degeneration, or toxic causes of parkinsonism.
* Patients with a cardiac pacemaker
* History of brain surgery or placement of a deep brain stimulator
* Psoriasis vulgaris (or other inflammatory skin condition) on or near skin where the vibro-acoustic device and sleep tracking ring will be donned.
* Patients on beta-blockers, benzodiazepines, antipsychotics, and stimulants (except for the treatment of attention deficit disorder/ADHD).
* Pregnancy
* Patients who begin cognitive behavioral therapy or a selective serotonin reuptake inhibitor (SSRI) medication for an anxiety disorder or other psychiatric disorder after the baseline clinical assessment.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-08-09 (Actual); Primary Completion 2023-08-09 (Actual); Study Completion 2023-08-09 (Actual)

PRIMARY OUTCOMES:
Average Nighttime Heart Rate Variability | after 90-120 days of intervention
  Average heart rate variability during the night, as measured by Oura ring device (measured in s).
Paced Auditory Serial Addition Test score | after 90-120 days of intervention
  A measure of cognitive function that assesses auditory information processing speed and flexibility, scored as the total number correct out of 60. Higher scores indicate better performance.
Spielberger State-Trait Anxiety Inventory score | after 90-120 days of intervention
  40-item questionnaire to assess anxiety. Scores range from 40-160 with higher scores indicating greater severity of anxiety.
Hamilton Anxiety Scale score | after 90-120 days of intervention
  14-item questionnaire to evaluate severity of anxiety symptoms. Scores range from 0-56, with higher scores indicating greater severity of anxiety.
Hamilton Depression Scale score | after 90-120 days of intervention
  17-item questionnaire to assess the severity of depression symptoms. Scores range from 0-61, with higher scores indicating more severe depression.
Beck Depression Inventory score | after 90-120 days of intervention
  21-item scale to evaluate the severity of depression symptoms. Scores range from 0-63, with higher scores indicating more severe depression.
Beck Anxiety Inventory score | after 90-120 days of intervention
  21-item questionnaire to assess the severity of anxiety. Scores range from 0-63, with higher scores indicating greater anxiety.
Geriatric Depression Scale score | after 90-120 days of intervention
  15-item questionnaire scored from 0-15, with greater scores indicating greater severity of depression.
Short Activities-specific Balance Confidence Scale score | after 90-120 days of intervention
  16-item scale to assess confidence in balance while performing different tasks. Scores range from 0-100 with greater scores indicating greater confidence.
New Freezing of Gait Questionnaire score | after 90-120 days of intervention
  9-item questionnaire evaluating the severity of freezing of gait. Scores range from 0-29, with higher scores indicating more severe freezing of gait.
Instrumental Activities of Daily Living Scale score | after 90-120 days of intervention
  8-item questionnaire to assess functional independence. Scores range from 0-8, with higher scores indicating higher functioning.
Insomnia Severity Index score | after 90-120 days of intervention
  7-item scale to assess severity of insomnia. Scores range from 0-28, with higher scores indicating greater severity of insomnia.
Epworth Sleepiness Scale score | after 90-120 days of intervention
  8-item scale to assess daytime sleepiness. Scores range from 0-24, with higher scores indicating greater daytime sleepiness.
Fatigue severity Scale score | after 90-120 days of intervention
  9-item scale to measure the severity of fatigue. Scores range from 9-63, with higher scores indicating greater severity of fatigue.
Perceived Stress Scale score | after 90-120 days of intervention
  10-item questionnaire to evaluate perceived levels of stress. Scores range from 0-40, with greater scores indicating greater perceived stress.
Short Fall Efficacy Scale International score | after 90-120 days of intervention
  7-item questionnaire to evaluate fear of falling. Scores range from 7-28 with greater scores indicating greater fear of falling.
Fatigue Visual Analogue Scale score (Alternate form) | after 90-120 days of intervention
  Scored from 0-100, with higher score indicating greater fatigue.
Mayo Sleep Questionnaire Score on item 8 | after 90-120 days of intervention
  Item 8 on the Mayo Sleep Questionnaire asks the participant to rate their general level of alertness over the past 3 weeks on a scale from 0 to 10, with 0 indicating they sleep all day and 10 indicating they are fully and normally awake.

CONTACTS AND LOCATIONS:
Overall Officials: Prabesh Kanel, PhD, Principal Investigator — University of Michigan
Locations (1):
- Domino's Farms, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No